CLINICAL TRIAL: NCT01867164
Title: A Prospective, Open-Label, Comparative, Parallel Double-Arm, Multicentric Clinical Study to Evaluate the Efficacy of an Ovule With Triple Active Agents (Terconazole, Clindamycin, Fluocinolone) Administered Once Per Day for Three Days Versus an Ovule With Triple Active Agents (Metronidazole, Nystatin, Fluocinolone) Administered Once Per Day for Ten Days to Treat Secondary Vulvar/Vaginal Symptoms of Vaginitis/Infectious Vaginosis (Bacterial and/or Mycotic and/or Parasitic)
Brief Title: A Study to Compare Efficacy and Safety of an Ovule Containing Terconazole, Clindamycin and Fluocinolone Versus an Ovule Containing Metronidazole, Nystatin and Fluocinolone in the Treatment of Secondary Vulvar/ or Vaginal Symptoms of Infectious Vaginitis/ and Infectious Vaginosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100569; TEROV8BAC4001
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-11

CONDITIONS: Vaginitis; Infectious Vaginosis
Keywords: Vaginitis; Infectious vaginosis; Terconazole; Clindamycin; Fluocinolone; Metronidazole; Nystatin
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gynoclin V (Experimental): One ovule containing 80 milligram (mg) terconazole, 100 mg clindamycin and 0.5 mg fluocinolone acetonide will be administered vaginally, every 24 hours at night, for 3 days.
  Interventions: Drug: Gynoclin V
- Vagitrol V (Experimental): One ovule containing 500 mg metronidazole, 0.5 mg fluocinolone acetonide and 100,000.00 microgram/milliliter nystatin will be administered vaginally, every 24 hours at night, for 10 days.
  Interventions: Drug: Vagitrol V

INTERVENTIONS:
Drug: Gynoclin V — One ovule containing 80 milligram (mg) terconazole, 100 mg clindamycin and 0.5 mg fluocinolone acetonide will be administered vaginally, every 24 hours at night, for 3 days.
  Arms: Gynoclin V
Drug: Vagitrol V — One ovule containing 500 mg metronidazole, 0.5 mg fluocinolone acetonide and 100,000.00 microgram/milliliter nystatin will be administered vaginally, every 24 hours at night, for 10 days.
  Arms: Vagitrol V

SUMMARY:
The purpose of this comparative study is to evaluate the efficacy of an ovule with triple active agents (terconazole, clindamycin and fluocinolone) versus another ovule with triple active agents (nystatin, metronidazole and fluocinolone) in the treatment of symptoms caused by the presence of vaginitis (inflammation of the vagina) or bacterial vaginosis (polymicrobial, nonspecific vaginitis associated with positive cultures of Gardnerella vaginalis and other anaerobic organisms and a decrease in lactobacilli).

DETAILED DESCRIPTION:
This is a prospective (study following participants forward in time), open-label (all people know the identity of the intervention), randomized (the study drug is assigned by chance), comparative, parallel (a clinical trial comparing the response in 2 or more groups of participants receiving different treatments) double-arm, multi-center (when more than 1 hospital or medical school team work on a medical research study) study. The study consists of 3 phases: Screening phase on Visit 1 (Day -3/1); Inclusion or treatment phase on Visit 2 (Day 1); and Treatment or monitoring phase (3 days after treatment) on Visit 3 (Day 7 for Gynoclin V and Day 13 for Vagitrol V) and Visit 4 (Day 12 for Gynoclin V and Day 18 for Vagitrol V). Participants will be randomly assigned to 1 of the 2 treatment groups: Gynoclin V and Vagitrol V. Participants in Gynoclin V group will be administered 1 ovule (containing 80 milligram [mg] terconazole, 100 mg clindamycin and 0.5 mg fluocinolone acetonide) vaginally every 24 hours at night, for 3 days. Participants in the Vagitrol V group will be administered 1 ovule (containing 500 mg metronidazole, 0.5 mg fluocinolone acetonide and 100,000.00 microgram/milliliter nystatin) vaginally every 24 hours at night, for 10 days. Primarily, participants will be evaluated for signs and symptoms, characteristics of vaginal discharge, changes in vulvar region, changes in cervix and presence of bacteria, fungi and/or parasites. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants presenting clinical symptoms compatible with vaginitis/bacterial vaginosis, with any of the following symptoms being the reason for the consultation: pruritus (itchiness), vulvar burning, as well as presenting leukorrhea (a clear or white discharge from the vagina, consisting mainly of mucus) as an accompanying symptom
* Participant who agrees to return at the 7th and 13th day after starting the treatment
* Participant who agrees to abstain from sexual relations for the 13 days of the study
* Participant who have signed informed consent to participate in the study

Exclusion Criteria:

* Participant with a known allergy to vaginal treatments
* Participants who have received treatment for the current condition in the 10 days before the date of inclusion, or is currently receiving antibiotics (drug used to stop or slow down the growth of germs), antifungals, anti-parasitics or systemic steroids
* Participant with suspected pregnancy or currently breastfeeding
* Participant who has received unknown drugs or experimental drugs within the 3 months before inclusion
* Participant known to be a carrier of a severe (very serious, life threatening) disease that alters the metabolism or excretion of the drugs used (liver or kidney disease)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A. Clinical Trial, Study Director — Janssen-Cilag, S.A.
Locations (2):
- Mexico (2):
  - DF, Mexico City
  - Mexico City

RESULTS

PARTICIPANT FLOW:
Groups:
- Gynoclin V (Terconazole+Clindamycin+Fluocinolone Acetonide): One ovule containing 80 milligram (mg) terconazole, 100 mg clindamycin and 0.5 mg fluocinolone acetonide was administered vaginally, every 24 hours at night, for 3 days.
- Vagitrol V (Metronidazole+Fluocinolone Acetonide+Nystatin): One ovule containing 500 mg metronidazole, 0.5 mg fluocinolone acetonide and 100,000.00 microgram/milliliter (mcg/ml) nystatin was administered vaginally, every 24 hours at night, for 10 days.
Period: Overall Study
Arm/Group | Gynoclin V (Terconazole+Clindamycin+Fluocinolone Acetonide) | Vagitrol V (Metronidazole+Fluocinolone Acetonide+Nystatin)
Started | 81 | 79
Completed | 81 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study medication and who were evaluated for efficacy parameters were included in Intent-to-treat (ITT) population.
Groups:
- Gynoclin V (Terconazole+Clindamycin+Fluocinolone Acetonide): One ovule containing 80 mg terconazole, 100 mg clindamycin and 0.5 mg fluocinolone acetonide was administered vaginally, every 24 hours at night, for 3 days.
- Vagitrol V (Metronidazole+Fluocinolone Acetonide+Nystatin): One ovule containing 500 mg metronidazole, 0.5 mg fluocinolone acetonide and 100,000.00 mcg/ml nystatin was administered vaginally, every 24 hours at night, for 10 days.
- Total: Total of all reporting groups
Arm/Group | Gynoclin V (Terconazole+Clindamycin+Fluocinolone Acetonide) | Vagitrol V (Metronidazole+Fluocinolone Acetonide+Nystatin) | Total
Number analyzed (Participants) | 81 | 79 | 160
Age Continuous [Mean (Standard Deviation); unit: Years] — Participants who received at least 1 dose of study medication and who were evaluated for efficacy parameters were included in ITT population. A total of 81 participants in Gynoclin V and 78 participants in Vagitrol V were analyzed for this Baseline characteristic.
  Years | 30.69 (7.17) | 30.56 (7.50) | 30.63 (7.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 79 | 160
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Presence or Absence of Symptoms 3 Days After Treatment
Description: Participants were evaluated for presence or absence of symptoms (itching, burning and sudden vulvar pain) in response to treatment.
Time Frame: 3 days after treatment (Day 7 for Gynoclin V or Day 13 for Vagitrol V)
Population: Participants who received at least 1 dose of study medication and who were evaluated for efficacy parameters were included in Intent-to-treat (ITT) population. Here 'N' specifies participants who were evaluated for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Gynoclin V (Terconazole+Clindamycin+Fluocinolone Acetonide) | Vagitrol V (Metronidazole+Fluocinolone Acetonide+Nystatin)
Number analyzed (Participants) | 79 | 77
Percentage of Participants
  Itching: Absent | 67.1 | 79.2
  Itching: Present | 32.9 | 20.8
  Burning: Absent | 78.5 | 88.3
  Burning: Present | 21.5 | 11.7
  Sudden vulvar pain: Absent | 95.0 | 90.9
  Sudden vulvar pain: Present | 5.0 | 9.1

2. Primary Outcome: Percentage of Participants With Presence or Absence of Symptoms 8 Days After Treatment
Description: as for outcome 1
Time Frame: 8 days after treatment (Day 12 for Gynoclin V or Day 18 for Vagitrol V)
Population: Participants who received at least 1 dose of study medication and who were evaluated for efficacy parameters were included in ITT population. Here 'N' specifies participants who were evaluated for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Gynoclin V (Terconazole+Clindamycin+Fluocinolone Acetonide) | Vagitrol V (Metronidazole+Fluocinolone Acetonide+Nystatin)
Number analyzed (Participants) | 77 | 75
Percentage of Participants
  Itching: Absent | 88.3 | 85.3
  Itching: Present | 11.7 | 14.7
  Burning: Absent | 93.5 | 92
  Burning: Present | 6.5 | 8
  Sudden vulvar pain: Absent | 97.4 | 89.3
  Sudden vulvar pain: Present | 2.6 | 10.7

3. Primary Outcome: Percentage of Participants With the Presence of Microorganisms (Single-celled, Tiny Organisms That Include Fungi, Bacteria, Viruses) 3 Days After Treatment
Description: Percentage of participants with the presence of microorganisms (Candida albicans, Candida species, Gardnerella vaginalis, Vaginal flora, Lactobacillus species) in the wet mount, KOH, gram stain and vaginal discharge culture (candida and symptomatology) 3 days after treatment.
Time Frame: 3 days after treatment (Day 7 for Gynoclin V or Day 13 for Vagitrol V)
Population: Participants who received at least 1 dose of study medication and who were evaluated for efficacy parameters were included in ITT population. Here 'N' signifies participants who were evaluated for this outcome measure including the participants for whom no culture was performed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Gynoclin V (Terconazole+Clindamycin+Fluocinolone Acetonide) | Vagitrol V (Metronidazole+Fluocinolone Acetonide+Nystatin)
Number analyzed (Participants) | 78 | 76
Percentage of Participants
  Candida albicans | 2.5 | 0
  Candida species, Gardnerella vaginalis | 9.8 | 1.3
  Vaginal Flora | 55.6 | 58.2
  Lactobacillus species | 28.4 | 36.7
  No culture performed | 3.7 | 3.8

4. Secondary Outcome: Percentage of Participants With Response to Treatment Assessed by Participant
Description: Response to treatment was evaluated by participant using a 5-point numerical scale: 1=No response (no improvement or condition even worsened); 2=Poor (No symptoms disappeared and symptoms are moderate to severe) 3=Moderate (improvement and symptoms are of moderate intensity); 4=Good (much improvement, but there are still some occasional mild symptoms); 5=Excellent (all symptoms disappeared).
Time Frame: 8 days after treatment (Day 12 for Gynoclin V or Day 18 for Vagitrol V)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Gynoclin V (Terconazole+Clindamycin+Fluocinolone Acetonide) | Vagitrol V (Metronidazole+Fluocinolone Acetonide+Nystatin)
Number analyzed (Participants) | 77 | 75
Percentage of Participants
  Poor | 1.30 | 1.30
  Moderate | 0 | 4.00
  Good | 36.40 | 29.40
  Excellent | 62.30 | 65.30

5. Secondary Outcome: Percentage of Participants With Response to Treatment Assessed by Physician
Description: Response to treatment was evaluated by Physician using a 5-point numerical scale: 1=No response (no improvement or condition even worsened); 2=Poor (No symptoms disappeared and symptoms are moderate to severe) 3=Moderate (improvement and symptoms are of moderate intensity); 4=Good (much improvement, but there are still some occasional mild symptoms); 5=Excellent (all symptoms disappeared).
Time Frame: 8 days after treatment (Day 12 for Gynoclin V or Day 18 for Vagitrol V)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Gynoclin V (Terconazole+Clindamycin+Fluocinolone Acetonide) | Vagitrol V (Metronidazole+Fluocinolone Acetonide+Nystatin)
Number analyzed (Participants) | 77 | 75
Percentage of Participants
  Poor | 1.30 | 1.30
  Moderate | 0 | 5.30
  Good | 28.60 | 26.70
  Excellent | 70.10 | 66.70

ADVERSE EVENTS:
Time Frame: Baseline up to Day 13 for Gynoclin V and Day 18 for Vagitrol V
Arm/Group | Gynoclin V (Terconazole+Clindamycin+Fluocinolone Acetonide) | Vagitrol V (Metronidazole+Fluocinolone Acetonide+Nystatin)
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/79
Other Adverse Events (participants affected / at risk) | 1/81 | 1/79
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gynoclin V (Terconazole+Clindamycin+Fluocinolone Acetonide) (N=81) | Vagitrol V (Metronidazole+Fluocinolone Acetonide+Nystatin) (N=79)
Fungal Infections (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No